CLINICAL TRIAL: NCT03763890
Title: Post- End- Expiratory Pressure Affect the Alveolar Heterogeneity in Moderate and Sever ARDS Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Director, Southeast University, China
Other Study IDs: 20181129PEEP
Record Dates: First submitted 2018-11-29; First posted 2018-12-04 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Ards
Keywords: ARDS（Acute respiratory syndrome）;; stress;; strain;; Trans-pulmonary pressure;; FRC(functional residual capacity ); PEEP（post end-expiratory pressure）;; EIT（Electronic impedance tomography）;; RVD(region ventilation delay)
MeSH Terms: conditions — Acute Lung Injury; Sprains and Strains

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Post-end-Expiratory pressure — Titrate the PEEP from 24 cmH2O to 6 cmH2O, 2 cmH2O/step and record EIT, trans-pulmonary pressure, hemodynamic parameter and Blood-gas analysis.

SUMMARY:
This study try to use EIT ( Electronic impedance tomography ) to evaluate the alveolar heterogeneity and use trans-pulmonary pressure and stain to evaluate the lung injury . The study use these methods to figure out how PEEP impact the alveolar heterogeneity and VILI.

DETAILED DESCRIPTION:
ARDS(Acute respiratory distress syndrome )is common in patients suffering Sepsis, trauma, burning and other sever condition and characterized by diffuse alveolar damage and alveolar heterogeneity.ARDS patient need MV(mechanical ventilation )to maintain oxygenation and need unique MV tragedy to avoid VILI(Ventilator induced Lung injury ).PEEP(post-end-expiratory pressure) is crucial to maintain oxygenation and avoid VILI according to researches. But there are also some other research different voice. This study try to use EIT ( Electronic impedance tomography ) to evaluate the alveolar heterogeneity and use trans-pulmonary pressure and stain to evaluate the lung injury . The study use these methods to figure out how PEEP impact the alveolar heterogeneity and VILI.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 or<80；
2. Moderate or sever ARDS in 2012 <Berlin definition>;
3. Applied mechanical ventilation;
4. Consent signed.

Exclusion Criteria:

1. Asthma or COPD；
2. Cardiogenic edema；
3. Sever neutropenia(<500/mm3)；
4. Hemodynamic astatic: DOPA or Dobutamine >15 µg/kg/ min; NE > 15ug /min；
5. GCS coma score ≤12；
6. Thoracic injury or surgery patients contradict EIT ；
7. Refuse to join in trail；
8. Included in other clinical trail。

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Moderate or sever ARDS in 2012 <Berlin definition>;
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
alveolar hyper-distention; alveolar collapse；alveolar opening and closing； | September,1,2018-December 30, 2020
  The study use Pulmo Vista 500 device (Drager co.),is intended to perform thoracic bioimpedance measurements by applying the technique of electrical impedance tomography (EIT)to evaluate alveolar hyper-distention(%of the lung volume); alveolar collapse(% of the lung volume)；alveolar opening and closing(% of the lung volume).
Trans-pulmonary pressure | September,1,2018-December 30, 2020
  The researchers place tube in the esophagus and connect it to transmitter to measure esophageal pressure (mmHg)and calculate trans-pulmonary pressure(mmHg) to evaluate stress
EELV | September,1,2018-December 30, 2020
  The research use nitrogen wash out to measure EELV（end-expiratory lung volume, ml） to calculate dynamic strain and evaluate the strain
peak pressure | September,1,2018-December 30, 2020
  The researchers use ventilator to measure peak pressure(cmH2O) in patients with mechanical ventilation and without spontaneous breathing..
plateau pressure | September,1,2018-December 30, 2020
  The researchers use ventilator to do inspiration pause to measure plateau pressure(cmH2O) in patients with mechanical ventilation and without spontaneous breathing.
tidal volume | September,1,2018-December 30, 2020
  The researchers use ventilator to measure tidal volume(ml) in patients with mechanical ventilation and without spontaneous breathing..
respiratory rate | September,1,2018-December 30, 2020
  The researchers record the set respiratory rate(bpm) in patients with mechanical ventilation.
flow | September,1,2018-December 30, 2020
  The researchers record the set Flow (L/min) in patients with mechanical ventilation.
FiO2 | September,1,2018-December 30, 2020
  The researchers record the set FiO2 ( fraction of inspiratory oxygen, %) in patients with mechanical ventilation.
PaO2 | September,1,2018-December 30, 2020
  The researchers use blood gas analysis to measure PaO2( arterial oxygen pressure,mmHg)
PaCO2 | September,1,2018-December 30, 2020
  The researchers use blood gas analysis to measure PaCO2( arterial carbon dioxide pressure,mmHg) .

SECONDARY OUTCOMES:
SBP | September,1,2018-December 30, 2020
  Recording SBP(systolic pressure, mmHg),which is always continuously monitored with invasive pressure monitor.
DBP | September,1,2018-December 30, 2020
  Recording DBP(Diastolic pressure, mmHg),which is always continuously monitored with invasive pressure monitor.
CVP | September,1,2018-December 30, 2020
  Recording CVP(central venous Pressure）,which is always discontinuously monitored with jugular pressure monitor mmHg).
vasopressor | September,1,2018-December 30, 2020
  Recording clinical vasopressor usage including Norepinephrine（ μg/Kg/min;）Epinephrine（μg/Kg/min） Dobutamine （ μg/Kg/min)

CONTACTS AND LOCATIONS:
Overall Officials: haibo qiu, PhD, Study Director — Nanjing Zhong-Da Hospital, Southeast University School of Medicine,China
Locations (1):
- Nanjing Zhong-Da Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No